CLINICAL TRIAL: NCT02325193
Title: Prevention of Hypoglycaemia Using the Minimed®640G System
Brief Title: "MiniMed 640G System" User Evaluation With the Question of Reducing the Rate of Hypoglycemia
Status: Completed | Type: Observational
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Collaborators: Medtronic International Trading Sarl (Industry)
Responsible Party: Principal Investigator, Thomas Danne, Prof. Dr. med., Kinderkrankenhaus auf der Bult
Other Study IDs: MM640G
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Minimed®640G system — Sensor augmented insulin therapy with and without use of Predictive low glucose management (PLGM)

SUMMARY:
The Minimed®640G system (MM640G) consists of a combination of insulin and glucose sensor for continuous glucose monitoring (CGM). Here, the glucose sensor transmits not only the continuous glucose data on the display of insulin pump but, in the case of hypoglycemia also interrupt their insulin delivery of pump. In the currently available system Paradigm®VEO, the interruption takes place at a settled threshold level. In difference in the new system MM640G the shutdown algorithm can already be proactive and help avoid hypoglycemia completely. The so called PLGM algorithm (predictive low glucose management) should be tested in the user evaluation. The main objective is to answer the question of reducing the rate of hypoglycemia by application of the new PLGM algorithm.

Included are a total of 24 patients, aged 1-21 years, in three pediatric diabetes centers.

DETAILED DESCRIPTION:
In the first phase of two weeks, the sensor-augmented pump therapy (SaP) is carried out without these interruption PLGM algorithm. In a second phase for 6 weeks, the PLGM function is set. Both phases are compared in terms of the rate of hypoglycemia, the time spent and the area under the curve (AUC) glucose range (values <70 mg / dl (3.9 mmol / l)).

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes, diagnosed since 12 month at least
* continuous subcutaneous insulin infusion (CSII) since 3 month at least
* stable outcome since 3 month at least
* willingness of patients/ parents to wear a glucose sensor for 2 month
* willingness of patients/ parents to use the Minimed®640G system
* willingness of patients/ parents to complete a diary
* willingness of patients/ parents to comply the requirements of the study protocol

Exclusion Criteria:

* longer absence of the patients (not able to attend the study visits)
* subject with allergy of sensor or specific sensor components
* communication problems
* significant history of eating disorder, anorexia, bulimia
* pregnancy
* significant history of drug abuse or/ and alcoholism
* patient do not want to attend the trial
* missing informed consent

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * patients with type 1 diabetes
  * CSII since 3 month at least
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
average AUC/day in hypoglycaemic range < 70mg/dl (3,9mmo/l) | 6 weeks

SECONDARY OUTCOMES:
Number of PLGM activities | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Danne, MD, Principal Investigator — Kinder - und Jugendkrankenhaus AUF DER BULT
Locations (1):
- Kinder - und Jugendkrankenhaus AUF DER BULT, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No